CLINICAL TRIAL: NCT00800982
Title: A Single-Center, Open-Label, Pilot Study to Evaluate the Efficacy and Tolerability of Narrow Band UVB Phototherapy in Enhancing Etanercept's Maintenance Dose in Obese Patients With Moderate to Severe Plaque-Type Psoriasis
Brief Title: Open Label Study Etanercept's Maintenance Dose in Obese Patients With Moderate to Severe Plaque Type Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOO - ENBREL-2008; H5939-31693-01 (Other: UCSF Committee for Human Research)
Record Dates: First submitted 2008-05-13; First posted 2008-12-03 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Psoriasis
Keywords: Obese patients (BMI>30); Patients with moderate to severe psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Etanercept only) (Active Comparator): Subjects will only be treated with etanercept. This is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months. No UVB will be given. Sham UVB will not be used because the subjects are not blinded because they often know they are receiving sham UVB due to differences in light intensity and heat.
  Interventions: Drug: etanercept
- 2 (Etanercept + nb-UVB) (Experimental): Subjects will receive etanercept. This is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months.
  In addition, for months 3-6, subjects will receive Narrow Band Ultraviolet B phototherapy three times a week for 12 weeks in addition to the etanercept maintenance dose. The safety and efficacy of the combination therapy will be evaluated by the registered phototherapy nurses at each phototherapy visit and by the study investigator at monthly visits. NB-UVB therapy will be adjusted according to the clinical judgment of the University of California San Francisco Psoriasis Treatment Center phototherapy staff.
  Interventions: Procedure: Narrow band (310-312 nm) ultraviolet light B phototherapy; Drug: etanercept

INTERVENTIONS:
Procedure: Narrow band (310-312 nm) ultraviolet light B phototherapy — Narrow band (310-312 nm) ultraviolet light B phototherapy 3 times a week during Weeks 12-24. NB-UVB therapy will be adjusted according to the clinical judgment of the University of California San Francisco Psoriasis Treatment Center phototherapy staff
  Other Names: nb-UVB; nbUVB; narrowband UVB
  Arms: 2 (Etanercept + nb-UVB)
Drug: etanercept — Etanercept is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months.
  Other Names: Enbrel

SUMMARY:
This is a single-center, open-label, pilot study. A total of 30 subjects (15 in each study arm) will be enrolled in this 6 month study to evaluate whether the addition of narrow band UVB (NB-UVB) phototherapy can enhance the efficacy of etanercept's maintenance dose, 50 mg once a week, in obese psoriasis patients.

DETAILED DESCRIPTION:
In Phase I, all subjects will receive etanercept's induction dose, 50 mg twice a week, for a total of 12 weeks. In Phase II, all subjects will receive etanercept's maintenance dose, 50 mg once a week, during Weeks 12-24. Those subjects randomized to the treatment arm will receive NB-UVB phototherapy 3 times a week during Phase II. In order to ensure homogeneity between the NB-UVB arm and non-NB-UVB arm, subjects will be randomized according to their Body Mass Index (BMI). The Psoriasis Area Severity Index (PASI) score and Physician Global Assessment (PGA) will be calculated at each visit to determine the effectiveness of the etanercept and NB-UVB treatment during both phases of the study. The hypothesis is that the combination of NB-UVB phototherapy three times a week and etanercept maintenance dose (50 mg once a week) will enhance the efficacy of the maintenance dose alone in obese patients (BMI >30) with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Nonimmunocompromised males or females 18 years of age or older.
* Must be able to read, understand, and speak basic English.
* Body Surface Area (BSA) involvement of greater than 10%.
* Psoriasis Area and Severity Index greater than 10.
* Obese defined as having a Body Mass Index greater than 30.
* Eligible for systemic therapy, particularly etanercept, and Narrow Band Ultraviolet B in the opinion of the investigator.
* Sign and date the appropriate written informed consent and Health Insurance Portability and Accountability Act authorization
* Negative urine pregnancy test within 7 days before the first dose of etanercept in all women (except those surgically sterile or at least 5 years postmenopausal).
* No evidence of active or latent tuberculosis based on a negative Purified Protein Derivative skin test. Patients with documentation of adequately treated tuberculosis may be enrolled.
* Sexually active subjects of childbearing potential must agree to use medically acceptable form of contraception during screening and throughout the study.
* Willing and able to self-administer subcutaneous injections or to have a qualified person available to administer subcutaneous injections
* Agrees to comply with protocol requirements, attend all regularly study visits and is considered to be a good study subject
* Meets concomitant medication washout requirements

Exclusion Criteria:

* Erythrodermic, pustular, or guttate psoriasis
* Evidence of skin conditions other than psoriasis that would interfere with study-related evaluations of psoriasis.
* Known sensitivity to any component of the study medications.
* Evidence of active infections such as fevers, chills, sweats, or history of untreated Lyme disease and active severe infections within 4 weeks before screening visit, or between the screening and Week 0 visits.
* Evidence of latent or active hepatitis B infection as indicated by positive HBsAg test during the screening visit.
* Personal or first degree family history of neurologic disease.
* Poorly controlled medical condition including, but not limited to, unstable cardiovascular disease, poorly controlled diabetes, recent stroke, history of recurrent infections, or any other condition for which, in the opinion of the investigator, participation in the study would place the subject at risk.
* History of any Tumor Necrosis Factor-α inhibitor use including etanercept, infliximab, and adalimumab within 4 weeks of starting study drug.
* History of non-cutaneous malignancy within the past 5 years.
* History of drug or alcohol abuse. Substance abuse must clearly be documented so those patients with a remote and minor history of drug/alcohol use will still have an opportunity to participate in the study.
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
* Plans to receive any live vaccines during the study.
* Evidence of photosensitivity disorder (i.e. polymorphous light eruption).
* Known photosensitivity or known sensitivity to any of the excipients or products to be administered during dosing.
* Current enrollment in another clinical study and treatment with another experimental drug or approved therapy for experimental use within 30 days prior to Week 0
* Cannot commit to all the assessments required by the protocol
* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Considered by the investigator, for any reason, to be an unsuitable candidate for study participation.
* Cannot or do not wish to comply with the protocol washout requirements (please see section below entitled "Washout Period Prior to Week 0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — UCSF Psoriasis and Skin Treatment Center, Department of Dermatology, University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States

REFERENCES:
- [Result] Park KK, Wu JJ, Koo J. A randomized, 'head-to-head' pilot study comparing the effects of etanercept monotherapy vs. etanercept and narrowband ultraviolet B (NB-UVB) phototherapy in obese psoriasis patients. J Eur Acad Dermatol Venereol. 2013 Jul;27(7):899-906. doi: 10.1111/j.1468-3083.2012.04611.x. Epub 2012 Jun 15. PMID 22702846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were July 2010 through June 2011. Recruitment was performed at the dermatologic medical clinic.
Pre-assignment Details: The following treatments for psoriasis required wash-out before group assignment: any type of ultraviolet B phototherapy or topical therapy for 14 days; psoralen and ultraviolet A or any oral or systemic psoriasis treatment for 28 days; alefacept or ustekinumab for 12 weeks, Tumor Necrosis Factor-a inhibitor or monoclonal antibody for 4 weeks.
Groups:
- 1 (Etanercept Only): Subjects will only be treated with etanercept. This is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months. No Ultraviolet B will be given. Sham Ultraviolet B will not be used because the subjects are not blinded because they often know they are receiving sham Ultraviolet B due to differences in light intensity and heat.
- 2 (Etanercept + Nb-UVB): Subjects will receive etanercept. This is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months.
  In addition, for months 3-6, subjects will receive Narrow Band Ultraviolet B phototherapy three times a week for 12 weeks in addition to the etanercept maintenance dose. The safety and efficacy of the combination therapy will be evaluated by the registered phototherapy nurses at each phototherapy visit and by the study investigator at monthly visits. Narrow Band Ultraviolet B therapy will be adjusted according to the clinical judgment of the University of California San Francisco Psoriasis Treatment Center phototherapy staff.
Period: Overall Study
Arm/Group | 1 (Etanercept Only) | 2 (Etanercept + Nb-UVB)
Started | 15 | 15
Completed | 13 | 12
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Patient moved out of state | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 (Etanercept + Nb-UVB): Subjects will receive etanercept. This is given at the standard FDA approved dosage of 50 mg twice weekly x 3 months then 50 mg once weekly x 3 months.
  In addition, for months 3-6, subjects will receive NB-UVB phototherapy three times a week for 12 weeks in addition to the etanercept maintenance dose. The safety and efficacy of the combination therapy will be evaluated by the registered phototherapy nurses at each phototherapy visit and by the study investigator at monthly visits. NB-UVB therapy will be adjusted according to the clinical judgment of the UCSF Psoriasis Treatment Center phototherapy staff.
- Total: Total of all reporting groups
Arm/Group | 1 (Etanercept Only) | 2 (Etanercept + Nb-UVB) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44.7 (1.8) | 43.8 (2.1) | 44.2 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area Severity Index. This Scale Ranges From 0-72, 0 Being no Disease, and 72 Being Most Severe. The Number of Patients Who Achieved 75% Improvement of Their Psoriasis at the End of 24 Weeks Are Indicated in the Outcomes Data Below.
Description: Psoriasis area severity index was used to determine the number of patients in each treatment arm who had 75% improvement in their psoriasis. This scale uses the characteristics of the psoriasis, such as body surface area, redness, thickness, and scaling, to determine the severity score.
Time Frame: Weeks 12-24
Population: All patients that completed the trial through week 24 were used for analysis.
Measure: Number; unit: participants
Arm/Group | 1 (Etanercept Only) | 2 (Etanercept + Nb-UVB)
Number analyzed (Participants) | 13 | 12
participants | 6 | 6

ADVERSE EVENTS:
Arm/Group | 1 (Etanercept Only) | 2 (Etanercept + Nb-UVB)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Of the 30 subjects enrolled, 3 were lost to follow-up, one moved out of state, and one voluntarily withdrew due to worsening of psoriasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No